CLINICAL TRIAL: NCT00597558
Title: Treatment of Egg Allergy in Children Through Oral Desensitization (EGG OIT)
Acronym: EggOIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2299
Record Dates: First submitted 2008-01-06; First posted 2008-01-18 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2017-01

CONDITIONS: Food Hypersensitivity
Keywords: Egg allergy
MeSH Terms: conditions — Food Hypersensitivity; Egg Hypersensitivity | interventions — Egg Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Egg white protein (Experimental): Subjects, who are egg allergic, are given egg white protein for desensitization with the hypothesis they will develop tolerance.
  Interventions: Drug: Egg white protein

INTERVENTIONS:
Drug: Egg white protein — Egg white protein powder
  Other Names: Egg OIT

SUMMARY:
The purpose of this study is to determine if children with egg allergy can be desensitized to egg protein and if this desensitization can help them outgrow their egg allergy at an earlier time than normal. Our hypothesis is that children with egg allergy can be orally desensitized to egg protein and that this desensitization will help them outgrow their egg allergy at an earlier time than normal.

DETAILED DESCRIPTION:
Egg allergy in children under 5 years of age is extremely common. Egg, along with milk and peanuts, cause 80% of the food allergy reactions in children in the United States. Children have allergic reactions to egg ranging from mild urticaria to systemic anaphylaxis. The current therapy for children with egg allergy is to place the child on an egg-free diet until the allergy is outgrown. Because egg protein is a part of a significant number of processed foods it is difficult to totally avoid all egg proteins. Accidental ingestions leading to reactions to egg can occur with a bite of a cookie (~70 mg of egg protein) or a bite of a cake (~55 mg of egg protein). Children typically do not outgrow their egg allergy for several years. Therefore it would be helpful if a specific form of therapy would make children outgrow their allergic reactions to egg sooner. Egg protein is given to children in this study in small increasing amounts to desensitize them to the egg protein with the goal of helping them to outgrow their allergy.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 to 16 years of age
* Diagnosed egg allergy by CAP FEIA to egg of 5 kU/l or greater (2 kU/l or greater if 2 years old or less) or have had a positive allergic reaction to egg within 6 months.
* Having eaten egg in his/her diet prior to diagnosis
* A family that will be able to be compliant with all study visits
* All females of child bearing age must be using appropriate birth control

Exclusion Criteria:

* History of anaphylaxis to egg
* Medical history that would prevent a DBPCFC (double-blind placebo-controlled food challenge) to egg. The medical history that would prevent the DBPCFC to egg would be a prior history of an open egg challenge in which the patient experienced hypotension which required fluid resuscitation, respiratory compromise which necessitated ventilatory support, or poorly controlled asthma as evidenced by an FEV1 < 80% of predicted, or FEV1/FVC <75%, with or without controller medications
* Unable to cooperate with challenge procedures or unable to be reached by telephone for follow-up
* Diagnosed corn allergy

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2003-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of Arkansas, Little Rock, Arkansas
  - UNC Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buchanan AD, Green TD, Jones SM, Scurlock AM, Christie L, Althage KA, Steele PH, Pons L, Helm RM, Lee LA, Burks AW. Egg oral immunotherapy in nonanaphylactic children with egg allergy. J Allergy Clin Immunol. 2007 Jan;119(1):199-205. doi: 10.1016/j.jaci.2006.09.016. Epub 2006 Oct 27. PMID 17208602
- [Result] Vickery BP, Pons L, Kulis M, Steele P, Jones SM, Burks AW. Individualized IgE-based dosing of egg oral immunotherapy and the development of tolerance. Ann Allergy Asthma Immunol. 2010 Dec;105(6):444-50. doi: 10.1016/j.anai.2010.09.030. PMID 21130382

RESULTS

PARTICIPANT FLOW:
Groups:
- Egg White Protein Powder: Egg allergic subjects who ingest oral egg white protein for desensitization and possible tolerance.
Period: Overall Study
Arm/Group | Egg White Protein Powder
Started | 13
Completed | 9
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Egg White Protein Powder
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 6.6 [3.6 to 13.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Double-blind, Placebo-controlled Food Challenge (DBPCFC) to Egg
Description: Subjects will have a double-blind, placebo-controlled food challenge (DBPCFC) to egg after at least 24 months of egg OIT when the IgE to egg is < 7 kU/L or 90% of entry level IgE or SPT <= 5mm with a maximum treatment period of 60 months.
Time Frame: 24-60 months
Measure: Number; unit: subjects with no symptoms on DBPCFC
Groups:
- Egg White Protein Powder: Egg allergic subjects who ingest oral egg white protein
Arm/Group | Egg White Protein Powder
Number analyzed (Participants) | 9
subjects with no symptoms on DBPCFC | 9

2. Secondary Outcome: Egg Protein Skin Prick Test After Egg OIT
Description: Wheal size on egg protein skin prick test at the end of egg OIT treatment compared with at baseline.
Time Frame: 24-60 months
Measure: Mean (Full Range); unit: mm
Arm/Group | Egg White Protein Powder
Number analyzed (Participants) | 9
mm | 1.8 [0 to 9]

3. Secondary Outcome: Serum CAP-FEIA to Egg
Description: Measure of serum CAP-FEIA to egg from subjects on egg OIT after completion of treatment compared to baseline
Time Frame: 24-60 months
Measure: Mean (Full Range); unit: ku/L
Arm/Group | Egg White Protein Powder
Number analyzed (Participants) | 9
ku/L | 4.7 [0.35 to 8.4]

ADVERSE EVENTS:
Time Frame: 24-60 months
Arm/Group | Egg White Protein Powder
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Egg White Protein Powder (N=13)
Erythematous rash (Skin and subcutaneous tissue disorders) | 6
Skin itch (Skin and subcutaneous tissue disorders) | 1
Hives (Skin and subcutaneous tissue disorders) | 3
Lip or eye swelling (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Nasal itch (Respiratory, thoracic and mediastinal disorders) | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal itch (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0
Eye itch (Eye disorders) | 1
Eye tearing (Eye disorders) | 0

LIMITATIONS AND CAVEATS:
Endpoints were based on reaching certain lab criteria and thus the time on treatment varied from 24-60 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No